CLINICAL TRIAL: NCT04512365
Title: Brain-Behavior Markers of Reward and Drug Effects in Young Adults
Brief Title: Reward and Drug Effects on Mood and Brain Response
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Natania A Crane, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-0189; 1K23DA048132-01A1 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cannabis Use; Healthy
Keywords: THC; adult
MeSH Terms: interventions — Glucose; Dronabinol

STUDY DESIGN:
Intervention Model Description: Half of the participants will receive placebo during the first laboratory visit and THC during the second laboratory visit. The other half of participants will receive THC during the first laboratory visit and placebo during the second laboratory visit.
Who Masked: Participant, Investigator
Masking Description: THC or placebo will be prescribed to participants by a licensed psychiatrist, and dispensed by the University of Illinois at Chicago's Investigational Drug Service (IDS). Staff at the Clinical Research Center will give the drug or placebo to participants with the PI or a physician designate, present on-site and/or available by pager.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo oral capsule (Placebo Comparator): Participants will receive a placebo at their first or second laboratory visit.
  Interventions: Drug: Placebo oral capsule
- THC (Experimental): Participants will receive THC (7.5 mg) at their first or second laboratory visit.
  Interventions: Drug: THC

INTERVENTIONS:
Drug: Placebo oral capsule — A capsule that contains only dextrose filler administered during the first or second laboratory visit.
  Other Names: Dextrose
  Arms: Placebo oral capsule
Drug: THC — A capsule that contains 7.5 mg of THC as well as dextrose filler administered during the first or second laboratory visit.
  Other Names: Marinol
  Arms: THC

SUMMARY:
The goal of the study is to better understand the neural mechanisms underlying the rewarding, reinforcing properties of delta-9-tetrahydrocannabinol (THC), the main psychoactive ingredient in cannabis, among healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* must be able to give informed consent
* age 18-25 at the time of signing the consent form
* fluency in English
* body mass index of 19-26 (normal/overweight but not obese due to limitations of MRI)
* negative urine drug screen (UDS) for all substances except THC (THC allowed)
* must be medically and neurologically healthy
* must not be taking psychoactive medications that would interfere with dronabinol and/or interpretation of fMRI data, including but not limited to the following classes of psychotropics: antidepressants, anxiolytics, sedative hypnotics, stimulants, antipsychotics, mood stabilizer
* have used cannabis at least 10 times in their life, but report current and past lifetime cannabis use less than 7 days/week (daily)

Exclusion Criteria:

* any current medical condition requiring psychoactive/psychotropic medication or medication that would interact with dronabinol, interpretation of fMRI data, and/or interfere with study procedures
* current or past allergic or adverse reaction or known sensitivity to cannabinoid-like substances (Dronabinol/Marijuana/Cannabis/THC, cannabinoid oil, sesame oil, gelatin, glycerin, and titanium dioxide.)
* current Axis-I Diagnostic Statistical Manual-5 diagnosis (although mild and moderate Cannabis Use Disorder (CUD) and mild and moderate Alcohol Use Disorder (AUD) are allowed)
* score >3 on the Prediction of Alcohol Withdrawal Severity Scale (PAWSS) for individuals with current AUD
* lifetime other lifetime Substance Use Disorder (although lifetime severe CUD and lifetime severe AUD are allowed)
* currently seeking or engaged in CUD treatment or have desire to cut down or stop cannabis use.
* in recovery or enrolled in treatment for any substance (including cannabis and alcohol)
* lifetime psychosis, mania, Attention-Deficit/Hyperactivity Disorder, Obsessive-Compulsive disorder, Feeding and Eating disorder, or Post-Traumatic Stress Disorder
* score >7 on the Hamilton Depression Rating Scale or score >7 on the Hamilton Anxiety Rating Scale
* less than a high school education
* lack of fluency in English
* night shift work
* currently pregnant confirmed by urine pregnancy test or planning pregnancy or lactating (women)
* unwilling/unable to sign informed consent document
* inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia), as determined by self-report
* left-handed
* presence of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
* positive UDS for any drug except THC
* positive breathalyzer for acute alcohol intoxication
* heavy alcohol use (>4 days week) in the past month
* heavy nicotine use (>20 cigarettes per week) in the past month

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Neural reward response- Reward Positivity (RewP) event-related potential | First and second laboratory visits, around 90 minutes to 2 hours after drug administration. Outcome measure is change from placebo session RewP to THC session RewP.
  Participants will complete the Doors task during electroencephalogram (EEG) capturing the RewP, with higher values indicating greater neural response to reward
Neural reward response- blood-oxygen-level-dependent (BOLD) response | First and second laboratory visits, around 90 minutes to 2 hours after drug administration. Outcome measure is change from placebo session BOLD response to THC session BOLD response.
  Participants will complete the Doors task during functional magnetic resonance imaging (fMRI) capturing BOLD response, with higher values indicating greater BOLD activation to reward
Subjective drug response- Addiction Research Center Inventory (ARCI)- Morphine Benzedrine Group (MBG) subscale | First and second laboratory visit, at baseline (Time 0) and at peak drug response (90-120 minutes) after drug administration. Outcome measure is change in peak score during placebo (peak minus baseline) compared to change in peak score during THC
  Participants will complete the ARCI-MBG self-report scale, with higher values reflecting more drug-induced euphoria

CONTACTS AND LOCATIONS:
Overall Officials: Natania A Crane, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No